CLINICAL TRIAL: NCT04992078
Title: A Prospective, Multi-Centre, Randomised Controlled Study to Evaluate the Clinical, Health Economic and Patient Reported Outcomes Following Unicompartmental Knee Arthroplasty With a Robotic Assisted Technique
Brief Title: A Comparison of Patients Receiving a Unicompartmental Knee Replacement With Robotic Assistance or With Conventional Instrumentation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been early terminated due to change of study protocol and study will be commence with new protocol and study number
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAVIO+JOURNEYUNI.2021.02
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Arthritis; Osteoarthritis; Knee; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
Keywords: Robotic; Unicompartmental Knee Replacement (UKR)
MeSH Terms: conditions — Arthritis; Osteoarthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Robotic-Unicompartmental Knee Replacement (R-UKR) (Experimental): NAVIO/CORI Surgical System
  Interventions: Device: NAVIO/CORI Surgical System
- Conventional-Unicompartmental Knee Replacement (C-UKR) (Active Comparator): Non-robotic conventional instrumentation
  Interventions: Procedure: Non-robotic conventional instrumentation

INTERVENTIONS:
Device: NAVIO/CORI Surgical System — Unicompartmental knee replacement with robotic assistance
  Arms: Robotic-Unicompartmental Knee Replacement (R-UKR)
Procedure: Non-robotic conventional instrumentation — Unicompartmental knee replacement with non-robotic conventional instrumentation
  Arms: Conventional-Unicompartmental Knee Replacement (C-UKR)

SUMMARY:
A unicompartmental (partial) knee replacement (UKR) is the removal of one part of the knee joint (a condyle), that has become damaged due to osteoarthritis, and replacing it with an artificial implant. The placement of these artificial implants and how they are aligned with each other is important because they can impact overall knee function and the long-term survival of the implant. A UKR is a highly effective, recognised procedure for patients with end-stage osteoarthritis affecting one compartment of the knee joint. The functional outcomes following UKA are at a minimum of equivalence to total knee arthroplasty procedures, with some recent literature demonstrating improved functional patient reported outcome scores.

There have been significant developments in knee replacement surgery over recent years. In particular, the introduction of robotic surgical systems, such as the NAVIO and CORI systems (Smith+Nephew Plc). These systems are hand-held devices which can support the surgeon with the knee replacement procedure, the systems are image-free and do not require the patient to undergo any scans (such as CT scans).

Comparisons of robotic systems to conventional instruments have demonstrated that robotic platforms produce fewer positioning errors in total knee replacement. This can result in more precise knee alignment and better outcomes following surgery. With both the NAVIO and CORI Surgical Systems there is a reduction in radiation exposure due to them being image-free.

At present, there is some evidence available for the long-term outcomes of knee replacement implanted using robotic assistance (i.e. 2-10 years) however this study is designed to look at the early outcomes following UKR. There is no literature to date to show that robotic-assisted UKR is superior to conventional methods, within the early post-operative period (up to 12 months).

This study is designed to show that the NAVIO/CORI surgical systems are better than conventional methods for UKR. The hypothesis is that they will be cost-effective, will reduce the time a patient spends in hospital following their surgery, will improve patient satisfaction during the early recovery period and will improve the patient's early post-operative mobility and function.

ELIGIBILITY:
Inclusion Criteria:

* Subject must provide written informed consent
* Subject must be aged 18 years or older at the time of surgery
* Subject is listed for a primary unicompartmental knee replacement (UKR)
* The indication for the UKR is primary arthritis of the knee joint involving one compartment
* The subject agrees to give informed consent to participate in the study including consenting to any incidental findings being reported to their General Practioner (GP)
* The subject agrees to consent to and to follow the study visit schedule
* The subject plans to be available throughout the 1-year post-operative period
* Routine radiographic assessment is possible

Exclusion Criteria:

* The subject undergoes a robotic-assisted UKR on the index joint as a revision for a previously failed surgery, or there is a need for complex implants, or any other implant than a standard unicompartmental knee arthroplasty (UKA)
* Subject is listed for a simultaneous bilateral UKR
* Subject does not understand written or spoken English used in the informed consent form
* Subject has active infection or sepsis
* Subject is to have a Smith+Nephew Journey II UNI implanted by non-robotic conventional instrumentation
* Subject is not available throughout the 1-year post-operative period
* Subject, in the opinion of the investigator, has a neuromuscular disorder that prohibits control of the index joint
* Subject is undergoing the surgery as a private patient
* Patients who, in the opinion of the clinical staff, do not have capacity to give consent
* Women who are pregnant
* Subjects with a medical or physical condition that, in the opinion of the investigator, would preclude safe subject participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Forgotten Joint Score (FJS) | Up to 1 year
  Subjects are asked to rate their awareness of their knee arthroplasty in 12 questions with a five-point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale with a high value reflecting the ability of the subject to forget about the replaced knee joint during the activities of daily living. The change from the baseline scores will be determined for each participant.

SECONDARY OUTCOMES:
Oxford Knee Score (OKS) | Up to 1-year post-operation
  The OKS contains 12 equally weighted questions on activities of daily living. Responses to each question range from 0-4 with a range of a possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome. The change from the baseline scores will be determined for each participant.
Oxford Arthroplasty Early Recovery Score (OARS) | Up to 6 weeks post-operation
  Subjects are asked to complete data regarding how they're feeling around four domains: Pain, Sleep, Nausea and feeling unwell, and Mobility. The OARS questionnaire is scored 0-100 with zero being a poor recovery and 100 being positive and indicative of a good recovery.
Oxford Arthroplasty Early Change Score (OACS) | Up to 6 weeks post-operation
  Subjects are asked to score how they feel after their surgery, compared to before, concentrating on areas such as ability, pain, overall feelings etc. The OACS questionnaire is scored from negative 50 to positive 50 with minus 50 being much worse than before surgery to 50 being much better than before surgery. Zero indicates no change from self-reported pre-operative health status.
Short-Form 12 Health Questionnaire (SF-12) | Up to 1-year post-operation
  The SF-12 is a health-related quality of life questionnaire consisting of 12 questions that measure eight health domains, taken from the original SF-36 questionnaire. The calculations of the Physical and Mental Health Composite scores produce a range of 0-100, a score of zero indicates the lowest level of health and 100 the highest level of health. The change from the baseline scores will be determined for each participant.
EuroQol Five-Dimensional Five-Level (EQ-5D-5L) | Up to 1-year post-operation
  The EQ-5D-5L is a health-related quality of life score comprising of 5 domains (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and the EQ Visual Analogue Scale (EQ-VAS). Patients are asked to rate their level of impairment across each of the domains. Health states are converted into a single index utility score using a scoring algorithm, a score of 1.0 indicates the best health state, lower scores indicate poorer health states. The change from the baseline scores will be determined for each participant.
EuroQol Visual Analogue Scale (EQ-VAS) | Up to 1-year post-operation
  The EQ-VAS provides a single global rating of self-perceived health, patients are asked to score their health on a scale of 0-100mm which represents the worst health they can imagine (a score of 0) and the best health they can imagine (a score of 100). The change from the baseline scores will be determined for each participant.
Visual Analogue Score (VAS)-PAIN | Up to 1-year post-operation
  Subjects will be asked to complete their pain levels on a scale of 0-100, 0 being no pain experienced and 100 meaning the worst pain possible. The change from the baseline scores will be determined for each participant.

OTHER OUTCOMES:
Timed Up and Go (TUG) Test | Up to 1-year post-operation
  The TUG test measures the time taken by the patient (in seconds) to rise from an armchair, walk 3 metres, turn round and return to sitting in the same chair, without physical assistance. The time taken to complete the test is strongly correlated to the level of functional mobility. The post-operative measurements will be compared to the baseline (pre-operative) time.
6-Minute Walk (6MW) Test | Up to 1-year post-operation
  The 6MW test measures the total distance walked in metres over a 6-minute duration, this test has been validated as a measure of functional performance following knee arthroplasty. The post-operative measurements will be compared to the baseline (pre-operative) distance.
Tibial Sagittal Alignment | Up to 1-year post-operation
  The tibial sagittal alignment (tibial slope) in degrees will be determined by measuring the angle between the tibial implant (bone interface) (or in the native knee the highest post between anterior and posterior aspects of tibia) and the tibial mechanical axis.
  The post-operative measurements will be compared to the baseline (pre-operative) measurements.
Femoral Sagittal Alignment | Up to 1-year post-operation
  The femoral sagittal alignment (flexion) in degrees will be calculated by measuring the angle between the femoral mechanical axis and the femoral implant axis on the box or pegs.
  The post-operative measurements will be compared to the baseline (pre-operative) measurements.
Coronal Alignment | Up to 1-year post-operation
  The femoral coronal alignment (MDFA) will be obtained by measuring the angle between the femoral mechanical axis and the medial to lateral axis of the condylar implant or femoral joint line.
  The tibial coronal alignment (MPTA) will be calculated by measuring the angle between the tibial mechanical axis and the medial to lateral axis of the tibial implant or tibial joint line.
  * *HKAA =MDFA + MPTA
  * *HKAA, hip-knee-ankle angle; MDFA, medial distal femoral angle; MPTA, medial proximal tibial angle
  The post-operative measurements will be compared to the baseline (pre-operative) measurements.
Mechanical Axis Alignment | Up to 1-year post-operation
  The mechanical axis alignment (MAA) will be measured from the long-leg radiographs and compared to the baseline (pre-operative) measurements.
  Alignment will be calculated using measurements taken through the centre of the hip (centre of the spherical femoral head), centre of the knee (centre of the tibial plateau) and centre of the ankle (centre of the talus).
Radiographic Assessment | Up to 1-year post-operation
  Radiographic assessment of the antero-posterior (A/P) and lateral (L) views shall be performed to identify the presence of radiolucent lines, osteolysis & implant migration.

CONTACTS AND LOCATIONS:
Overall Officials: Iain McNamara, Principal Investigator — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK)
Locations (6):
- Kilcreene Regional Orthopaedic Hospital, Kilkenny, Ireland
- United Kingdom (5):
  - Royal Orthopaedic Hospital, Birmingham, West Midlands
  - Edinburgh Royal Infirmary, Edinburgh
  - Central Middlesex Hospital, London
  - St Mary's Hospital, London
  - Norfolk and Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: No